CLINICAL TRIAL: NCT05774886
Title: Pilot Study of an Implantable Microdevice to Evaluate Drug Responses in Situ in Early-stage Triple-negative Breast Cancer
Brief Title: Implantable Microdevice for TNBC - Pilot Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: On hold
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ana C Garrido-Castro, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-508
Record Dates: First submitted 2023-01-31; First posted 2023-03-20 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Triple Negative Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer; Early Stage Triple-Negative Breast Carcinoma; Breast Neoplasms; Breast Carcinoma
Keywords: Triple Negative Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer; Early Stage Triple-Negative Breast Carcinoma; Breast Neoplasms; Breast carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- IMD Placement and Retrieval (Experimental): * Participants with confirmed anatomic stage II-III TNBC whose planned treatment includes neoadjuvant systemic therapy with the intention to undergo surgery, including breast and/or axillary surgery, will be selected for study participation.
  * Participants will undergo image-guided placement of 2 microdevices within a single lesion.
  * Participants will undergo image-guided retrieval of the microdevices (and surrounding tissue) approximately 72 hours after placement.
  * Participants will be monitored for safety endpoints and clinical data will be collected for the duration of the study.
  Interventions: Combination Product: Implantable Microdevice (IMD)

INTERVENTIONS:
Combination Product: Implantable Microdevice (IMD) — * Small, implantable device with 30 reservoirs for drug and drug combinations.
  * Placement of 2 microdevices into tumor will be performed via needle, percutaneously, and guided by interventional radiologic techniques.
  * Drugs include all or a subset of the following: Doxorubicin, Paclitaxel, Carboplatin, Eribulin, Pembrolizumab, Atezolizumab, Tazemetostat, Panobinostat, Olaparib, Capecitabine, Sacituzumab govitecan, Abemaciclib, Venetoclax, Doxorubicin + cyclophosphamide (combination), Doxorubicin + cyclophosphamide + paclitaxel + carboplatin (combination), Carboplatin + paclitaxel (combination), Doxorubicin + cyclophosphamide + pembrolizumab (combination), Doxorubicin + cyclophosphamide + paclitaxel + carboplatin + Pembrolizumab (combination), Paclitaxel + atezolizumab (combination), Paclitaxel + pembrolizumab (combination), Carboplatin + gemcitabine + pembrolizumab (combination), Carboplatin + paclitaxel + pembrolizumab (combination), Trastuzumab deruxtecan

SUMMARY:
The goal of this research study is to evaluate the safety and feasibility of implanting and retrieving a microdevice that releases microdoses of a specific drug or combination of drugs as a possible tool to evaluate the effectiveness of several cancer drugs against early stage Triple Negative Breast Cancer (TNBC).

The name of the intervention involved in this study is:

Implantable Microdevice (IMD)

DETAILED DESCRIPTION:
This is a single-arm, pilot research study to evaluate the safety and feasibility of using an implantable microdevice to measure local intratumoral response to chemotherapy and other clinically relevant drugs in triple-negative breast cancer (TNBC). A pilot study means that this is the first time investigators are examining this study intervention in TNBC. Participants selected for this study must have a diagnosis of Stage II-III TNBC and are scheduled to undergo neoadjuvant systemic therapy.

This study involves implanting 2 microdevices, each small enough to fit inside the tip of a needle, into a tumor. The microdevices will release microdoses of up to 30 different cancer drugs via passive diffusion. The drugs will only penetrate the local tumor tissues. After approximately 72 hours, the microdevices and small regions of surrounding tissue will be removed and studied.

The U.S. Food and Drug Administration (FDA) has not approved the microdevice as treatment for any disease. For this study, the drugs used are agents approved by the U.S. FDA for the treatment of different types of cancer.

The research study procedures include screening for eligibility, study treatment with evaluations, radiology scans of tumors, blood tests, tumor biopsies, mammograms, and follow-up visits.

It is expected that about 24 people will take part in this research study.

Participants will be followed on this study for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer.
* Anatomic stage II-III breast cancer per AJCC 8th edition classification system. Primary breast tumor must be at least 2 cm in size (per imaging and/or physical exam). Participants must be considered candidates for neoadjuvant systemic therapy with the intention to undergo surgery (breast +/- axillary).
* Estrogen-receptor and progesterone-receptor expression both <10% by immunohistochemistry (IHC), and HER2-negative status as determined by the current ASCO/CAP guidelines.
* Participant must agree to undergo the percutaneous procedures for implantation and removal of the microdevice.
* Participant must be evaluated by a surgeon and/or medical oncologist who will determine the clinically appropriate treatment strategy based on clinical history and extent of disease. Participant must be deemed medically fit to undergo the percutaneous procedures for microdevice implantation and removal.
* Participant must have a primary breast tumor that is considered amenable to percutaneous placement and removal of the microdevice. Participants with history of prior malignancy (invasive or in situ) in the ipsilateral breast are not eligible.
* Patients with multifocal or multicentric disease are eligible, if not known to be HER2-positive. Pathologic confirmation of multifocal or multicentric is at physician´s discretion; however, if pathologic confirmation is obtained, receptor status must be available prior to registration.
* Patients with bilateral breast cancers are eligible, if not known to be HER2-positive. Pathologic confirmation of bilateral breast cancer is at physician´s discretion; however, if pathologic confirmation is obtained, receptor status must be available prior to registration.
* Prior systemic therapy: No prior chemotherapy, biologic therapy, hormonal therapy or investigational therapy for this breast cancer.
* Prior radiation therapy: No prior radiation to the ipsilateral breast.
* Prior surgery: No prior surgery to the ipsilateral breast.
* The subject is ≥ 18 years old.
* ECOG performance status ≤ 2 (Appendix A).
* Participants will undergo laboratory testing within 7 days prior to the microdevice placement. Participants must have normal coagulation and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 75,000/mcL
  * PT (INR) < 1.5
  * PTT < 1.5 x control
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior registration. Childbearing potential is defined as: participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus).
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled, significant intercurrent or recent illness including, but not limited to, ongoing or active infection, uncontrolled non-malignant systemic disease, uncontrolled seizures, or psychiatric illness/social situation that would limit compliance with study requirements in the opinion of the treating investigator.
* Prior hypersensitivity to any of the study drugs implanted with the device.
* Pregnant women are excluded from this study because of the possible increased dose of radiation from imaging associated with the device placement (e.g., if placement cannot be performed guided by ultrasound or MRI, if additional imaging and/or procedures are required due to potential complication of the device placement or removal).
* Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or percutaneous biopsy procedures.
* Significant risk factors (including, but not limited to, high risk of venous thrombosis, pulmonary embolism, stroke, or myocardial infarction) precluding the safe cessation of anticoagulation medication as per Radiology guidelines. (Patients taking low-dose aspirin only do not need to be excluded.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | up to 80 hours
  Defined by assessment of adverse events as defined by CTCAE v5.0.
Number of Participants with Successful Procedure | up to 80 hours
  Defined as the ability to retrieve two implanted microdevices with sufficient tissue, of sufficient quality, for downstream histopathology analysis and interpretation of at least 67% of the microdevice reservoirs in each device.

SECONDARY OUTCOMES:
Local Intratumoral Response (per Apoptosis) | up to 80 hours
  Descriptive statistics will be used to summarize the quantitative measurement of apoptosis (apoptotic index) for drug-treated regions compared to untreated regions of the device.
Local Intratumoral Response (per Proliferation) | up to 80 hours
  Descriptive statistics will be used to summarize the quantitative measurement of proliferation (Ki67) for drug-treated regions compared to untreated regions of the device.
Response to Systemic Neoadjuvant Therapy (RCB Class) | up to 3 years
  Correlation between local intratumoral response with the microdevice and response to systemic neoadjuvant therapy will be evaluated. Clinical response to systemic neoadjuvant therapy will be defined using residual cancer burden (RCB) class.
Response to Systemic Neoadjuvant Therapy (RCB Score) | up to 3 years
  Correlation between local intratumoral response with the microdevice and response to systemic neoadjuvant therapy will be evaluated. Clinical response to systemic neoadjuvant therapy will be defined using RCB score.
Invasive disease-free survival | up to 3 years
  Correlation between local intratumoral response with the microdevice and invasive disease-free survival, defined as the time from registration until the occurrence of local/regional recurrence, contralateral invasive breast cancer, distant recurrence, second primary invasive non-breast cancer, or death due to any cause or censored at date of last disease evaluation.
Overall survival | up to 3 years
  Correlation between local intratumoral response with the microdevice and overall survival, defined as the time from registration until death due to any cause or censored at the date of last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Garrido-Castro, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu